A study to evaluate the efficiency of trans-perineal trigger point dry needling combined with manual therapy as a treatment for chronic pelvic pain compared with treatment by manual therapy only: An open-label clinical trial.

NCT0279502

Version date: 28/08/2018



**Clinical Research Ethics Committee of the Cork Teaching Hospitals.** 

**Study Protocol** 

Aim

The presence of myofascial trigger points (MTrPs) or tender points in the pelvic floor

muscles (PFM) can attribute to myofascial pelvic pain (MFPP). MFPP is considered to be a

cause for chronic pelvic pain (CPP) symptoms including dyspareunia. This study will

evaluate the efficiency of including trans-perineal trigger point dry needling (TrDN) with

manual therapy to target MTrPs in the PFM compared to manual therapy alone.

The primary objective is to evaluate the number of treatments required within the allocated

ten treatment sessions to effect improvement in pain in the treatment groups.

**Preface** 

The aetiology of CPP can originate from urological, gynaecological, gastrointestinal, pelvic

neural and pelvic musculoskeletal systems (1,2,3). Non-cyclical CPP does not present

exclusively with symptoms of dyspareunia, dyschezia or dysuria. It can present with

additional symptoms such as suprapubic and lower abdominal pain, and painful pelvic

musculatures (2). The pain can worsen after pelvic floor related activities such as coitus or

voiding (4). Furthermore, non-cyclical CPP can also present with worsening of dysmenorrhea

symptoms due to hormonal changes, giving a mixed cyclical presentation without the

presence of an underlying gynaecological pathology (1).

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

Due to overlapping symptoms found in cyclical-CPP and non-cyclical CPP and the potential

presence of an underlying pathology, a multi-disciplinary approach to diagnosis and

management is crucial (1,5). Only 60% of laparoscopic investigations yield a definite

diagnosis (6). An inconclusive diagnosis with no evident pathology should suggest

myofascial pelvic pain (MFPP) as a probable cause (7). MFPP is caused by the presence of

MTrPs in the pelvic muscles, and its presence in PFM can be the primary mediator for non-

cyclical CPP (7,8).

Preface to treatments for MFPP

Manual therapy

Empirically, trigger point release (TPR) or myofascial tender point release (MFR) and

massage have been standard treatments for MTrPs in myofascial pain syndromes (MPS) (9).

Manual therapy for CPP symptoms such as Interstitial cystitis/ Painful Bladder Syndrome

(IC/PBS), vulvodynia and dyspareunia have been proved useful (10-14). These studies

reviewed manual techniques used externally for abdominal and pelvic muscles as well as

intra-vaginal and intra-rectal procedures for the PFM. These procedures varied from TPR,

global therapeutic massage (GTM), distension of shortened muscles and ligaments either

manually or with a therapeutic glass wand (TW).

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

**Trigger point dry needling** 

Trigger point dry needling (TrDN) is a minimally invasive treatment, where an acupuncture

needle is inserted directly into the muscle to target the underlying MTrPs, to change the

biochemical milieu and reduce neuromuscular pain and dysfunction (15). It is also considered

as an intra-muscular technique to increase the range of movement (ROM) of the muscles due

to the direct intramuscular stretch effect with the insertion of a needle (16).

Literature review on treatment sessions required to assess improvement with manual

therapy

Five randomised clinical trials (RCT) analysed manual therapy with treatment-based

interventions (12,13,14,17,18) and had a clinically significant resolution of pain and

dyspareunia at follow-up but required ten to twelve treatments for the duration of six months.

The number of treatments required for improvement in pain was analysed in only one RCT

(17). This study (17) compared the outcomes of Levator Ani trigger point injection (LTPI) of

local anaesthesia to manual therapy for pelvic floor pain. The treatment duration for

improvement in the physiotherapy group (n= 17) was over 7.3 weeks with resolution seen in

35% of the group compared to 81% achieving pain resolution in 4.4 weeks in the injection

group (n= 12). This study found that with increased manual treatments, the pain with

intercourse domain on the Female Sexual Function Index (FSFI) questionnaire for the

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

physiotherapy group showed more significant improvement (p=0.02), from a baseline of 1.74

to 4.14 compared to the injection group's statistics of 2.80 to 3.60 (17). This indicates that

treatment techniques that restore length in the muscles rather than therapies targeting pain

alone would be more efficacious.

The RCT (12) comparing myofascial release of the PFM with global therapeutic massage for

PBS suffering participants; found that 59% (n= 38) in the physiotherapy group showed a

marked improvement with ten treatments compared to only 26% (n=40) in the GTM group

(p=0.0012).

One of the first cohort studies (10) to evaluate the benefits of intra-vaginal TPR of muscles

for PBS and overactive bladder syndrome achieved 83% marked improvement with 24

sessions.

A pilot RCT (14) (n=9) reviewed the efficacy of self-release of tender points using a

therapeutic wand and found twice the improvement in bladder pain when myofascial self-

release of the PFM was continued and extended as a home exercise program for six weeks

after the cessation of six weeks of physiotherapy treatments.

Heyman et al. (13) compared stretching of the PFM (n=22) to counselling for dyspareunia.

This is the only study that showed an improvement in the pelvic pain scores for the distention

group (p<0.001) with fewer sessions of four to six treatments.

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

These studies (10,12,14,17) showed the relevance of manual therapy for PFM but required

over ten sessions for the observed improvement. The stand-alone efficiency of manual

treatments for pelvic floor pain and tightness is unclear as some studies have investigated the

outcome of physiotherapy alongside medical or psychological interventions and required

eight sessions extending from eight to 24 weeks to show significant improvement (18-20).

Literature review on treatment sessions required with dry needling

In a physiotherapy practice, TrDN is used in conjunction with manual therapy, stretching and

exercises. There is evidence that TrDN is an effective treatment to target MTrPs causing

MPS (21-24). A systematic review (24) on low back pain (LBP), showed that TrDN when

combined with physiotherapy treatments, had a more significant effect in pain improvement

with a lower visual analogue scale (VAS) of 1.04cms score than the treatments alone. The

treatment duration for the four intervention-based studies varied from 20 days to nine weeks.

The review (22) on TrDN for upper-body MPS analysed one study comparing TrDN

combined with shoulder rehabilitation. A more significant decrease in pain was noted for the

TrDN group with a minimal clinically important difference (MCID) of 1.81cms on the VAS

when TrDN was administered four times every five to seven days.

In a meta-analysis (23), the study that included TrDN with stretches showed a significant

increase in the ROM of the muscles (p=0.043) compared to stretches alone. The treatment

duration was three weeks.

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

An RCT (25) that reviewed stretches combined with TrDN for chronic non-specific neck pain

found 58% (n=65) in the combined intervention group required only two treatments from the

allocated four to report resolution of symptoms.

A study (26) on temporomandibular dysfunction (TMD) found that the deep TrDN technique

for MTrPs (n=36) had a lasting effect for up to six months post-treatment and showed a

significant improvement in pain and increased ROM of the jaw after just one treatment for

three weeks (p<0.01).

**Research Hypotheses** 

Null hypothesis: The inclusion of trans-perineal TrDN to manual therapy will not influence

the number of treatments required to achieve a clinically meaningful reduction in pain within

the allocated ten sessions. It will not affect the outcomes for the pain variables and

dyspareunia across the categories of treatments.

Research hypothesis: The inclusion of trans-perineal TrDN to manual therapy will influence

the number of treatments required to achieve a clinically meaningful reduction in pain within

the allocated ten sessions along with a variation in outcomes across the variables evaluated.

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

Method

This open label non-randomised clinical trial will compare two interventions pre-and post-

treatment. This trial will be analysed by intention to treat. The ethical approval was obtained

from the Clinical Research Ethics Committee of the Cork Teaching Hospitals in March 2016.

The trial is conducted at the Cork University Maternity Hospital (CUMH) and the Cork

Women's Clinic (CWC). CUMH is a large Obstetrics and Gynaecology hospital governed by

the Health Service Executive. CWC is a private gynaecology clinic. Female participants will

be referred for physiotherapy as deemed appropriate by the inclusion and exclusion criteria

(Table 1) given to the gynaecology team at CUMH and CWC.

The primary objective is to evaluate the number of treatments required within the allocated

ten treatments to effect improvement in pain in both groups. Pain resolution will be assessed

using the 0-10 Numeric Pain Rating Scale (0-10 NPRS). NPRS will be given at baseline, the

fourth, the eighth and the tenth treatment or earlier if resolution of symptoms occurred

without the requirement of the allocated ten treatments. The secondary objective is to

compare the outcomes between the treatment arms for dyspareunia, bladder and

musculoskeletal pain, and some menstrual cycle related pain symptoms with the Female

Sexual Function Index questionnaire and an abbreviated version of the International Pelvic

Pain Questionnaire (IPPQ). These questionnaires will be completed at pre-treatment and at

the final session. The Pain Treatment Satisfaction Scale questionnaire (PTSS) measures the

treatment satisfaction in both groups which will be provided only at the final treatment.

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

### Table 1: Inclusion and exclusion criteria for recruitment

#### **Inclusion criteria**

- Females with non-cyclical CPP including dyspareunia and associated pelvic floor pain-related dysfunctions such as bladder pain, pain with urination or dyschezia.
- They should present with palpable high pelvic floor muscle tone and tenderness on vaginal examination in a clinical setting with a pain score of >4/10.
- They can present with lower abdominal pain, pelvic pain and/or groin pain and pain on sitting.
- Pain worsened with pelvic floor stretching activities like insertion of tampon or intercourse (27).
- Visceral conditions like interstitial cystitis are difficult to exclude at gynaecology review, as they can mimic CPP symptoms (1).
- Smokers are included.
- Nulliparous and parous women included.
- Age 18 to 60 years

#### **Exclusion criteria**

- Body mass index greater than 30, as the required needle length is not available.
- Chronic back pain of over 6 month duration and under pain management team.
- Orthopaedic back surgeries with implants.
- Pelvic pathologies like endometriosis, fibroids, cysts and polycystic ovarian syndrome.
- Pregnancy related pelvic girdle pain.
- Pregnant during the trial.
- Pelvic organ carcinomas.
- Undergoing cancer treatment.
- After gynaecology surgery of less than 16 weeks.
- After cardiovascular, gastroenterology, renal or orthopaedic surgery of less than 6 month's postoperative.
- Neurological conditions such as stroke, epilepsy, Parkinson's disease etc.
- Fibromyalgia and chronic fatigue syndrome.
- Undergoing any treatment such as Botox or analgesic injections which can interfere with physiotherapy outcomes.

## Exclusion criteria for dry needling

- Extreme needle phobia, rheumatoid arthritis, prolonged corticosteroid treatment, warfarin treatment, heart implants and blood clotting disorders.
- Participant should have no significant learning disability and should be able to understand the procedure to consent for a vaginal examination and for treatment.
- Participant should not require a chaperone during treatment in order to avoid administrative issues.

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

Recruitment and allocation

Women will be invited for the trial with a letter of invitation. On confirmation of interest in

the trial, their medical record numbers and names will be documented onto an excel sheet

with the month of referral. In order to accommodate for the CUMH physiotherapy waiting

list and to allow for the clinical workings at CUMH, an excel sheet with six names will be

emailed to the central appointments office at CUMH. Two CUMH secretaries unrelated to the

trial will randomly allocate the names into two opaque envelopes marked as group A and

group B.

The staff will allocate appointments for group A among three Chartered Physiotherapists in

Women's Health and Continence involved in the trial, including the researcher. The

participating physiotherapists will have no input in the allocation process and they all have

clinical experience of over 15 years.

Group B will be treated only by the researcher who has a clinical experience of eight years

using trans-perineal TrDN. An identical procedure will be piloted at the CWC. The

researcher will provide the treatment for both groups at the CWC. The participant's file will

be marked as Group A or B to inform about allocation. The recruitment process will ran from

April 2016 to November 2017.

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

Withdrawal from participation

An individual can decline participation in the trial at any stage of the trial. If a participant

reports needle phobia after group allocation, she will be transferred to group A. If a

participant refuses dry needling treatment after starting the treatment in group B, she will be

removed from the trial but care will continue.

**Interventions** 

**Group A: Manual therapy** 

The assessment includes a musculoskeletal assessment for pelvic anatomy and the pelvic and

abdominal muscles. The PFM tone will be reviewed with a vaginal and/or rectal assessment

(27, 28). The treatment consisted of myofascial TPR of MTrPs in the abdominal, pelvic and

pelvic floor muscles and the appropriate stretching for the required muscles. If symptoms

included lumbo-pelvic symptoms (27, 29), TPR and stretches for the lumbo-pelvic area will

be provided. As a cohort of heterogeneous symptoms is expected to be recruited, an HEP of

stretches for the muscles is to be prescribed as per the clinicians' judgement.

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

**Group B: Trans-perineal TrDN with manual therapy** 

Group B will receive an identical assessment as group A. The treatment consists of the

addition of trans-perineal dry needling for the PFM and TrDN for the pelvic and the

abdominal muscles. The HEP for group B will be prescribed as per the clinician's judgement.

Manual therapy is utilised in pelvic floor areas difficult to access with acupuncture needles.

With pelvic floor hypertonicity, pelvic floor contractions are painful and difficult to initiate

and the PFM is slow to return to the normal vaginal resting tone (VRT). Performing a few

contractions during vaginal assessment can help assess hypertonicity and tightness in the

PFM however, Kegel's based pelvic floor muscle training (PFMT) is contraindicated as they

can increase pain and hypertonicity and hence PFMT was not advised (7 p.8). The HEP for

both groups are lengthening exercises for the PFM assisted with diaphragmatic breathing.

Diaphragmatic breathing is influenced and altered by MFPP. An altered breathing pattern can

influence the VRT, where the woman guards and holds her PFM with an apical inspiration

instead of using a diaphragmatic inspiration to normalise the VRT. Re-education on the

breathing patterns is considered as an important HEP for both groups to help prevent

guarding and increasing the VRT. (30 p.333-334, 31,32).

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

Standardisation of assessment

Standardised assessment for both groups will be as follows

1. Subjective assessment

2. Gynaecological evaluation of PFM

- Dermatome and myotome examination

- Intra-vaginal identification of PFM as per Haslam J et al. (28)

- Muscle status (28)

3. Criterions for MTrPs identification in the pelvic muscles and the PFM (33)

- The muscle should elicits tenderness on palpation

- Pain reproduced on palpation of an MTrP in the muscle

- Pain reproduced in the referred zone on palpation, i.e., the area of complaint.

4. Standardized assessment for the lumbo-pelvic region if required

The European Guidelines standardised tests for the diagnosis of pelvic girdle pain are to be used if indicated in a non-aetiology specific presentation of CPP symptoms (34). The tests are

as follows:

- Distraction sacroiliac joint pain provocation test

- Posterior pelvic pain provocation test

- Long dorsal ligament test

- Active straight leg raise test

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

A positive test finding in any of the above tests requires further assessment for pelvic muscle tenderness (3). Pelvic-related pain patterns are to be evaluated based on Table 2.

**Table 2: Pelvic muscle related pain patterns** (3,7,35,36)

| Pelvic-pain patterns | Muscles involved |
|---|---|
| Suprapubic pain | 1.Illio-psoas 2.Lower quadrant abdominal muscles (7) 3.PFM (36) |
| Groin pain | 1.Adductor group of muscles 2.Lower quadrant abdominal muscles (7) 3. Pectineus 4. PFM (3) |
| Posterior pelvic pain | 1.Gluteal muscles 2. Illio-psoas (7) 3.Piriformis 4. QL (35) |
| Deep pelvic pain | 1.Adductor group of muscles 2. PFM (7) |

**Clinical Research Ethics Committee of the Cork Teaching Hospitals.** 

Standardisation of interventions

Standardisation of interventions is only required for group A as three clinicians provided the

treatment for this group. Physiotherapists specialising in gynaecology have in-depth

knowledge about intra-vaginal PFM palpation. For assessment, the PFM is divided into the

superficial PFM and the deep PFM. To access MTrPs and perform TPR in the individual

PFM, palpation varies based on the depth and the bulk of a muscle. On identification, manual

pressure of a recommended two kilograms (36) is to be applied to activate the MTrP, while

keeping the patient's tolerance in consideration. The pressure varies from five seconds up to

60 seconds based on the individual's tolerance or when the spontaneous pain generated eases

to a comfortable level. A rest period of 15 to 60 seconds is recommended between each TPR

(37). The treatment can last from 30 to 45 minutes depending on the number of muscles

involved. Tables 3.1 and 3.2 provides the procedure, frequency and treatment for group A

and B.

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

Table 3.1: Procedure, treatment and frequency for group A

# Procedure **Treatment and Frequency** Group A: 1<sup>st</sup> treatment – Trial checklist to be completed by Initial assessment of posture, spine and the the physiotherapist. PFM. Treatment is for 30-45 minutes on consent for treatment. Assess and treat with Consent forms to be filled by the participants. manual therapy for the PFM, pelvic and Complete three baseline questionnaires (NPRS, abdominal muscles if indicated. FSFI, IPPQ). **Frequency** – The treatment is scheduled for Subjective and objective assessment along with every two weeks unless the participant has her education of muscle involvement and treatment menstrual cycle or due to personal issues. The entailed. Education on good bladder, bowel and appointment was then rescheduled for the week dietary habits if indicated. Signing of consent after. forms for treatment and the trial. Assess and treat The HEP are stretches for the pelvic musculature with TPR and distention for the PFM, pelvic and as per presentation of CPP pain patterns. The abdominal muscles as per presentation. patient is advised the application of cryotherapy 4<sup>th</sup> treatment – complete NPRS for 15 minutes if she was sore after treatment. 8<sup>th</sup> treatment-complete NPRS 10<sup>th</sup> treatment or when ceasing treatments due **to positive outcomes** – to complete four final questionnaires (NPRS, FSFI, IPPQ, PTSS). 10<sup>th</sup> treatments – if no resolution is achieved, complete the final questionnaires and discharge from the trial but care continues.

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

Table 3.2: Procedure, treatment and frequency for group B

# Procedure

## Group B:

1<sup>st</sup> treatment – Trial check list to be completed by the physiotherapist. Consent forms to be filled by the participants.

Complete three baseline questionnaires (NPRS, FSFI, IPPQ).

Subjective and objective assessment along with education of pelvic muscle involvement and treatment entailed. Education on good bladder, bowel and dietary habits if indicated. Signing of consent forms for treatment, TrDN and trial.

Assess and treat with TrDN, TPR and distention for the PFM, pelvic and abdominal muscles per presentation.

4<sup>th</sup> treatment – complete NPRS

8<sup>th</sup> treatment-complete NPRS

10<sup>th</sup> treatment or final treatment- due to positive outcomes, complete four final questionnaires (NPRS, FSFI, IPPQ, PTSS).

10<sup>th</sup> treatments – if no resolution is achieved, complete the final questionnaires and discharge from the trial but care continues.

## **Treatment and Frequency**

Initial assessment of posture, spine and PFM.

Treatment is for 30-45 on consent for treatment.

Only introduce TrDN if the participant is happy to start treatment.

2<sup>nd</sup> treatment- To perform superficial TrDN technique for the PFM as an introduction to the deep needling technique if the patient is apprehensive about TrDN followed by compression and stretching of the PFM. If the participant is particularly nervous, start with needling muscles that are segmentally-related to the PFM such as the piriformis, rectus abdominous, gluteus and adductors.

For trans-perineal TrDN for the PFM, start with needling the Levator-ani muscles followed by the required deep PFM and then if required needle the superficial PFM. The patient is advised application of cryotherapy for 15 minutes if sore after treatment.

Frequency- Identical to group A.

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

Statistical analysis and power calculation

Since this is the first study to analyse TrDN for the PFM, the power in these studies

(12,13,25) were compared and it was estimated that in order to determine a p < 0.05, with 80%

power,  $\alpha$ =0.05,  $\beta$ =0.2, SD=1 for the outcome in the population and an effect size of 0.634, a

total of 80 participants will be required. One hundred and twenty four participants will be

invited as a participation rate of 70% is expected. Since studies analysing manual

interventions for pelvic floor pain were not statistically significant (12,13), MCID was

considered to be of practical significance. In chronic pain management, a 50% decrease in

pain from baseline is rated as significant improvement, while a 30% decrease is rated as a

meaningful improvement (38). Statistical analysis will be carried out using the IBM corp.

SPSS software 24. Visual inspection of Histograms and Q-Q plots will be utilised to check

the distribution of variables. A General Linear Model will be used to determine if the groups

differed with regard to mean pain level at the endpoint of the study with pre-treatment score

as the covariate in the analysis. The Kaplan Meier, non-parametric tests and Related Sample

Wilcoxon Signed rank test are to be used for between-groups and within-group analysis.

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

**Data monitoring** 

All questionnaires will be filled by the participants prior to their session at CUMH, CWC or

at their homes. The data will be stored in secure locked storage at the Physiotherapy

department at CUMH. The data collection will be undertaken by the researcher and a

physiotherapist unrelated to the trial. On completion of the trial, the data will analysed for

correct input by two doctors and one physiotherapist at CUMH who will be appointed as the

data monitoring committee. An interim analysis will not be conducted for this trial.

**Trial Duration:** 

The trial aims to run for two years.

**Clinical Research Ethics Committee of the Cork Teaching Hospitals.** 

### References

- 1. Daniels JP, Khan KS. Chronic pelvic pain in women. *BMJ* . 2010; 341:c4834–c4834.Available from: http://www.bmj.com/cgi/doi/10.1136/bmj.c4834.
- 2. Moore J, Kennedy S. Causes of chronic pelvic pain. *Best Practice & Research Clinical Obstetrics & Gynaecology*. 2000; 14:3:89–402.
- 3. Tu FF, As-Sanie S, Steege JF. Prevalence of pelvic musculoskeletal disorders in a female chronic pelvic pain clinic. *The Journal of Reproductive Medicine*. 2006; 15; p. 185–9. Available from: http://www.ncbi.nlm.nih.gov/pubmed/16674013
- 4. Butrick CW. Pelvic Floor Hypertonic Disorders: Identification and Management.

  Obstetrics and Gynecology Clinics of North America. 2009; 36: p. 707–22.
- Fall M, Baranowski AP, Elneil S, Engeler D, Hughes J, Messelink EJ, et al. EAU guidelines on chronic pelvic pain. *European Urology*. 2010; 57(1):35–48. Available from: http://www.sciencedirect.com/science/article/pii/S0302283809008604
- 6. Porpora MG, Gomel V. The role of laparoscopy in the management of pelvic pain in women of reproductive age. *Fertility and Sterility*. 1997; 68(5): p. 765–79.
- 7. Pastore EA, Katzman WB. Recognizing myofascial pelvic pain in the female patient with chronic pelvic pain. *Journal of Obstetrics Gynecology& Neonatal Nursing*. 2012; 41(5):680–91. https://doi.org/10.1111/j.1552-6909.2012.01404.x
- 8. Faubion SS, Shuster LT, Bharucha AE. Recognition and management of nonrelaxing

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

Ref no: EMC 4 (kk) 01/03/16 & EMC 3(jj) 04/04/17.

- pelvic floor dysfunction. Mayo Clinic Proceedings. Elsevier Inc. 2012; 87(2):187-93.
- 9. Travell JG, Simons DG. Myofascial Pain and Dysfunction: In: Williams & Wilkins (eds.): *The Trigger Point Manual*. Volumen 1.1983.
- 10. Weiss JM. Pelvic floor myofascial trigger points: manual therapy for interstitial cystitis and the urgency-frequency syndrome. *The Journal of Urology*. 2001; 166(6):2226–31. Available from: http://www.ncbi.nlm.nih.gov/pubmed/11696740
- 11. Anderson RU, Harvey RH, Wise D, Nevin Smith J, Nathanson BH, Sawyer T.
  Chronic Pelvic Pain Syndrome: Reduction of Medication Use After Pelvic Floor Physical
  Therapy with an Internal Myofascial Trigger Point Wand. *Applied Psychophysiologiy Biofeedback.* 2015; 40(1):45–52.
- 12. Fitzgerald MP, Payne CK, Lukacz ES, Yang CC, Peters KM, Chai TC, et al. Randomized multicenter clinical trial of myofascial physical therapy in women with interstitial cystitis/painful bladder syndrome and pelvic floor tenderness. *The Journal of Urology*. 2012; 187(6):2113–8. https://doi.org/10.1016/j.juro.2012.01.123
- 13. Heyman J, Ohrvik J, Leppert J. Distension of painful structures in the treatment for chronic pelvic pain in women. *Acta Obstetricia et Gynecologica Scandinavica*. 2006; 85(5):599–603.
- 14. Bond J, Pape H& Ayra CA. Efficacy of a therapeutic wand in addition to physiotherapy for treating bladder pain syndrome in women: a pilot randomized controlled trial. *Journal of Pelvic, Obstetrics Gynaecology Physiotherapy.* 2017; 120:12–27. Available from:

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

Ref no: EMC 4 (kk) 01/03/16 & EMC 3(jj) 04/04/17.

http://hdl.handle.net/10454/12129

- 15. Dommerholt J, Mayoral del Moral O, Gröbli C,Sandalcidi D, Langevin HM,. Trigger Point Dry Needling. *Journal of Manual & Manipulative Therapy*. Elsevier; 2006; 14(4):70E–87E. [Accessed 2017 Feb 4]. Available from: http://www.thedryneedlinginstitute.net/wp-content/uploads/2012/02/Myofascial-Dry-Needling.pdf
- Jafri MS. Mechanisms of Myofascial Pain. *International Scholarly Research Notices*.
   2014; 2014:1–16. Available from: http://www.hindawi.com/journals/isrn/2014/523924/
- 17. Zoorob D, South M, Karram M, Sroga J, Maxwell R, Shah A, et al. A pilot randomized trial of levator injections versus physical therapy for treatment of pelvic floor myalgia and sexual pain. *International Urogynecology Journal*. 2015; 26(6):845–52.

https://doi.org/10.1007/s00192-014-2606-4

- 18. Goldfinger C, Pukall CF, Thibault-Gagnon S, McLean L, Chamberlain S. Effectiveness of Cognitive-Behavioral Therapy and Physical Therapy for Provoked Vestibulodynia: A Randomized Pilot Study. *The Journal of Sexual Medicine*. 2016; 13(1):88–94. https://doi.org/10.1016j.jsxm.2015.12.03
- 19. Bergeron S, Binik YM, Khalife S, Pagidas K, Glazer HI, Meana M. A randomized comparison of group cognitive--behavioral therapy, surface electromyographic biofeedback, and vestibulectomy in the treatment of dyspareunia resulting from vulvar vestibulitis. *Pain*. 2001; 91. Available from: http://dx.doi.org/10.1016/S0304-

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

- 20. Bergeron S, Khalife S, Dupuis M-J, McDuff P. A randomized clinical trial comparing group cognitive-behavioral therapy and a topical steroid for women with dyspareunia. *Journal of Consulting and Clinical Psychology*. 2016; 84(3):259–68.
- 21. Tough EA, White AR, Cummings TM, Richards SH, Campbell JL. Acupuncture and dry needling in the management of myofascial trigger point pain: A systematic review and meta-analysis of randomised controlled trials. *European Journal of Pain. European Federation of Chapters of the International Association for the Study of Pain*; 2009; 13(1):3–10. Available from: http://dx.doi.org/10.1016/j.ejpain.2008.02.006
- 22. Kietrys DM, Palombaro KM, Azzaretto E, Hubler R, Schaller B, Schlussel JM, et al. Effectiveness of Dry Needling for Upper Quarter Myofascial Pain: A Systematic Review and Meta-Analysis. *Journal of Orthopedic & Sports Physical Therapy* . 2013; 43(9):1–46. doi: 10.2519/jospt.2013.4668
- 23. Rodriguez-Mansilla J, Gonzalez-Sanchez B, De Toro Garcia A, Valera-Donoso E, Garrido-Ardila EM, Jimenez-Palomares M, et al. Effectiveness of dry needling on reducing pain intensity in patients with myofascial pain syndrome: a Meta-analysis. *Journal of Traditional Chinese Medicine*. 2016; 36(1):1–13.

https://doi.org/10.1016/S0254-6272(16)30001-2

24. Liu L, Huang Q-M, Liu Q-G, Thitham N, Li L-H, Ma Y-T, et al. Evidence for Dry Needling in the Management of Myofascial Trigger Points Associated with Low Back

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

Pain: A Systematic Review and Meta-analysis. *Archives of Physical Medicine and Rehabilitation*. 2018; 99(1):144-152. Available from: http://linkinghub.elsevier.com/retrieve/pii/S0003999317304525

- 25. Cerezo-Téllez E, Torres-Lacomba M, Fuentes-Gallardo I, Perez-Muñoz M, Mayoral-Del-Moral O, Lluch-Girbés E, et al. Effectiveness of dry needling for chronic nonspecific neck pain: a randomized, single-blinded, clinical trial. *Pain* . 2016; 157(9):1905–17.

  Available from: http://www.ncbi.nlm.nih.gov/pubmed/27537209
- 26. Gonzalez-Perez LM, Infante-Cossio P, Granados-Nuñez M, Urresti- Lopez FJ. Treatment of temporomandibular myofascial pain with deep dry needling. *Medicine Oral, Patologia Oral Y Cirugia Bucal.* 2012; Sep 17(5):e781-785. doi:10.4317/medoral.17822 http://dx.doi.org/doi:10.4317/medoral.17822
- 27. Quaghebeur J, Wyndaele J-J. Chronic pelvic pain syndrome: Role of a thorough clinical assessment. *Scandinavian Journal of Urology* . 2015;49(2):81–9. Available from: http://www.tandfonline.com/doi/full/10.3109/21681805.2014.961546
- 28. J. Haslam & J. Laycock. Ever increasing circles. *Journal of Association of Chartered Physiotherapists in Women's Health*. 2009; 104:27–33.
- 29. Stuge B, Morkved S, Haug Dahl H, Vφllestad N. Abdominal and pelvic floor muscle function in women with and without long lasting pelvic girdle pain. *Manual Therapy*. 2006; 11(4):287–96. <a href="https://doi.org/10.1016/j.math.2005.07.003">https://doi.org/10.1016/j.math.2005.07.003</a>
- 30. Chaitow L. Chronic pelvic pain: Pelvic floor problems, sacro-iliac dysfunction and the

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

Ref no: EMC 4 (kk) 01/03/16 & EMC 3(jj) 04/04/17.

- trigger point connection. *Journal of Bodywork and Movement Therapy*. 2007; 11(4):327-339. https://doi.org/10.1016/j.jbmt.2007.05.002
- 31. Whelan Maeve CL. Practical anatomy, examination, palpation and manual release technique for the pelvic floor. In: *Chronic pelvic pain and dysfunction: Practical Physical Medicine*. Elsevier Churchill Livingstone; 2012. p. 311.
- 32. Hanno PM, Burks DA, Clemens JQ, Dmochowski RR, Erickson D, Fitzgerald MP, et al. AUA guideline for the diagnosis and treatment of interstitial cystitis/bladder pain syndrome. *The Journal of Urology*. 2011; 185(6):2162-2170.

  https://doi.org/10.1016/j.juro.2011.03.064
- 33. Gerwin RD, Shannon S, Hong CZ, Hubbard D, Gevirtz R. Interrater reliability in myofascial trigger point examination. *Pain*. 1997; 69:65–73. https://doi.org/10.1016/S0304-3959(96)03248-4
- 34. Vleeming A, Albert HB, Östgaard HC, Sturesson B, Stuge B. European guidelines for the diagnosis and treatment of pelvic girdle pain. *European Spine Journal*. 2008; 17: 794–819. https://doi.org/10.1007/s00586-008-0602-4
- 35. Torstensson T, Butler S, Lindgren A, Peterson M, Eriksson M, Kristiansson P. Referred pain patterns provoked on intra-pelvic structures among women with and without chronic pelvic pain: A descriptive study. *PLOS ONE*. 2015; 10(3). Available from: http://dx.doi.org/10.1371/journal.pone.0119542
- 36. Sanses TVD, Chelimsky G, McCabe NP, Zolnoun D, Janata J, Elston R, et al. The Pelvis

Clinical Research Ethics Committee of the Cork Teaching Hospitals.

Ref no: EMC 4 (kk) 01/03/16 & EMC 3(jj) 04/04/17.

and Beyond: Musculoskeletal Tender Points in Women With Chronic Pelvic Pain.

\*Clinical Journal of Pain. 2016;32(8):659–65. Available from:

http://www.ncbi.nlm.nih.gov/pubmed/26491938%0Ahttp://www.pubmedcentral.nih.gov/articlerender.fcgi?artid=PMC4840091

- 37. Fernández-De-Las-Peñas C, Alonso-Blanco C, Fernández-Carnero J, Carlos Miangolarra-Page J. The immediate effect of ischemic compression technique and transverse friction massage on tenderness of active and latent myofascial trigger points: A pilot study.

  Journal of Bodywork and Movement Therapy. 2006; 10(1):3–9.

  <a href="https://doi.org/10.1016/j.jbmt.2005.05.003">https://doi.org/10.1016/j.jbmt.2005.05.003</a>
- 38. Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, et al.

  Interpreting the Clinical Importance of Treatment Outcomes in Chronic Pain Clinical

  Trials: IMMPACT Recommendations. *Journal of Pain*. 2008;9(2):105–21.

  https://doi.org/10.1016/j.jpain.2007.09.005

Clinical Research Ethics Committee of the Cork Teaching Hospitals.